CLINICAL TRIAL: NCT04384991
Title: A Multicenter, Randomized, Double Blind, Restasis-controlled Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of HU007 Eye Drops in Patients With Dry Eye Syndrome
Brief Title: HU007 Eye Drops in Patients With Dry Eye Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Huons Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HU-007_P3-1
Record Dates: First submitted 2019-08-16; First posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HU007 Eye drop (Experimental): Adminster twice a day(one drop would be administered to both eyes once a time). When being administered, the IP should be mixed by upside down.
  Medication is recommended at 9AM(±1H) and 9PM(±1H)
  Interventions: Drug: HU007
- Restasis Eye drop 0.05% (Cyclosporine) (Active Comparator): Adminster twice a day(one drop would be administered to both eyes once a time). When being administered, the IP should be mixed by upside down.
  Medication is recommended at 9AM(±1H) and 9PM(±1H)
  Interventions: Drug: Restasis eye drop

INTERVENTIONS:
Drug: HU007 — Cyclosporine 0.02% with Trehalose 3%
  Arms: HU007 Eye drop
Drug: Restasis eye drop — Cyclosporine 0.05%
  Arms: Restasis Eye drop 0.05% (Cyclosporine)

SUMMARY:
This study is a multicenter, randomized, double blind, Restasis-controlled non-inferiority, Phase III Study to evaluate the efficacy and safety of HU007 eye drops in patients With dry eye syndrome

ELIGIBILITY:
Inclusion Criteria:

* Male and Female who over 19 years old
* Those who meet below criteria at least one of two eyes

  1. Those who have over than score 2 in corneal staining test-Oxford grading
  2. Tear secretion test without anesthesia(Schirmer test) result would be under 10mm/5min (If the test result is 0mm/5min, it should be over than 3mm/5min on the nasal stimulation schirmer test in the same eye)
  3. TBUT(Tear film break-up time) test result should be under 10sec.
* Woman with no possibility of pregnancy or negative pregnancy test results at a screening visit, Women or men who have agreed to maintain at least one contraceptive method during study period
* Those who could understand this study and agree to informed consent voluntarily

Exclusion Criteria:

* Those who have clinically significant eye disease not related to dry eye symdrome
* Those who are in anti-inflammatory medication for dry eye syndrome
* Medication of systemic steroid or immunosuppressant
* Those who have worn contact lenses before 72hours or have to wear contact lenses or disagree not to wear contact lenses during study period
* Those who have medical history with intraocular surgery 90 days before screening visit
* Those who have any active ophthalmic diseases such as active allergy, anterior uveitis, stevens-johnson syndrom which could affect the surfece of eye
* Those who have any autoimmune diseases
* Those who need a surgery for surface elevation caused by meibomian gland dysfunction(MGD)
* Those who have any medical history of corneal transplantation or neurotrophic keratitis
* Those who have diagnosed with glaucoma or have an intraocular pressure over than 25mmHg at least in one of the eyes
* Those who have medicated cyclosporine or steroid eye-drops 30 days before screening visit
* Those who have underwent any eye correction surgery such as LASIK(Laser-assistant in situ keratomileusis) 12 months before screening visit
* Those who have underwent a silicone lacrimal punctal occlusion or cauterization of the punctum excluding collagen lacrimal punctal occlusion 90 days before screening visit
* Those who have a hypersensitivity reaction for cyclosporine, trehalose or protein-based medication related to investigational drug
* Those who have diagnosed a psychical disorder which could affect this study
* Women who is pregnant or breastfeeding or those who have a plan to be pregnant
* Those who have medical history on abusing medications or alchol
* Those who have received other investigational drugs/devices 30 days before screening visit
* Those who are inappropriate for participating in this study according to investigator's judgement

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2019-05-03 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2019-12-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in corneal staining score-Oxford grading | Week 12
  Change from baseline in corneal staining score-Oxford grading at Week 12

SECONDARY OUTCOMES:
Change from baseline in corneal staining score-Oxford grading | Week 4, 8
  Change from baseline in corneal staining score-Oxford grading at Week 4, 8
Change from baseline in conjunctival staining score-Oxford grading | Week 4, 8, 12
  Change from baseline in conjunctival staining score-Oxford grading at Week 4, 8, 12
Change from baseline in strip meniscometry | Week 4, 8, 12
  Change from baseline in strip meniscometry at Week 4, 8, 12
Change from baseline in Tear film break-up time | at Week 4, 8, 12
  Change from baseline in Tear film break-up time at Week 4, 8, 12
Change from Baseline of Standard patient evaluation of eye dryness questionnaire | at Week 4, 8, 12
  Change from Baseline of Standard patient evaluation of eye dryness questionnaire at Week 4, 8, 12
Time to achieve 100% clearance on the corneal staining score | upto week 12
  Time to achieve 100% clearance on the corneal staining score

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, South Korea

IPD SHARING:
Plan to Share IPD: No
IPD would be substituted for screening or random No.